CLINICAL TRIAL: NCT02952534
Title: TRITON2: A Multicenter, Open-label Phase 2 Study of Rucaparib in Patients With Metastatic Castration-resistant Prostate Cancer Associated With Homologous Recombination Deficiency
Brief Title: A Study of Rucaparib in Patients With Metastatic Castration-resistant Prostate Cancer and Homologous Recombination Gene Deficiency
Acronym: TRITON2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: pharmaand GmbH (Industry)
Collaborators: Foundation Medicine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO-338-052; 2016-003162-13 (EudraCT Number)
Record Dates: First submitted 2016-10-24; First posted 2016-11-02 (Estimated); Results first posted 2022-06-08 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
Keywords: CRPC; PARP inhibitor; PARPi; BRCA; ATM; HRD; TRITON; homologous recombination; DNA repair; DNA defect; DNA anomaly; BARD1; BRIP1; CDK12; CHEK2; FANCA; NBN; PALB2; RAD51; RAD51B; RAD51C; RAD51D; RAD54L; germline; somatic; mCRPC
MeSH Terms: conditions — Mental Retardation, X-Linked, With Or Without Seizures, Arx-Related | interventions — rucaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rucaparib (Experimental): Oral rucaparib (monotherapy)
  Interventions: Drug: Rucaparib

INTERVENTIONS:
Drug: Rucaparib — Rucaparib will be administered daily
  Other Names: CO-338

SUMMARY:
The purpose of this study is to determine how patients with metastatic castration-resistant prostate cancer, and evidence of a homologous recombination gene deficiency, respond to treatment with rucaparib.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years old at the time the informed consent form is signed
* Have a histologically or cytologically confirmed adenocarcinoma or poorly differentiated carcinoma of the prostate
* Be surgically or medically castrated, with serum testosterone levels of ≤ 50 ng/dL (1.73 nM)
* Experienced disease progression after having received at least 1 but no more than 2 prior next-generation androgen receptor-targeted therapies, and 1 prior taxane-based chemotherapy, for castration-resistant disease
* Have a deleterious mutation in BRCA1/2 or ATM, or molecular evidence of other homologous recombination deficiency

Exclusion Criteria:

* Active second malignancy, with the exception of curatively treated non-melanoma skin cancer, carcinoma in situ, or superficial bladder cancer
* Prior treatment with any PARP inhibitor, mitoxantrone, cyclophosphamide or any platinum-based chemotherapy
* Symptomatic and/or untreated central nervous system metastases
* Pre-existing duodenal stent and/or any gastrointestinal disorder or defect that would, in the opinion of the investigator, interfere with absorption of rucaparib

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2021-07-18 (Actual); Study Completion 2021-07-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (149):
- United States (58):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinc, Phoenix, Arizona
  - Arizona Oncology Associates, Tucson, Arizona
  - Alliance Research Centers, Laguna Hills, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Sharp Memorial Hospital, San Diego, California
  - Pacific Hematology Oncology Associates, San Francisco, California
  - San Francisco VA Health Care System, San Francisco, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Redwood Regional Medical Group, Santa Rosa, California
  - Kaiser Permanente Medical Center (Vallejo), Vallejo, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - 4701 Ogletown Stanton Rd., Newark, Delaware
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Boca Raton Community Hospital, Inc., Boca Raton, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - University of Florida Health Cancer Center, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Atlanta Urological Group, Atlanta, Georgia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Ochsner Medical Center, New Orleans, Louisiana
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Walter Reed Hospital, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Fairview Hospital, Edina, Minnesota
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Minnesota Veterans Research Institute, Minneapolis, Minnesota
  - HCA Midwest Division - Kansas City, Kansas City, Missouri
  - Alegent Health Bergan Mercy Hospital , GU Research Network, Omaha, Nebraska
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Premier Urology Associates dba/AdvanceMed Research, Lawrenceville, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park, Buffalo, New York
  - NYU Perlmutter Cancer Center, New York, New York
  - Memorial Sloan Kettering CC, New York, New York
  - Weill Cornell Medical College/NewYork-Presbyterian Hospital, New York, New York
  - Premier Medical Group of the Hudson Valley PC, Poughkeepsie, New York
  - University of Rochester, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Carolina Urology Partners, Concord, North Carolina
  - The Urology Group, Cincinnati, Ohio
  - Kettering Cancer Center, Kettering, Ohio
  - Clinical Research Solutions, Middleburg Heights, Ohio
  - VA Portland Health Care System, Portland, Oregon
  - Consultants in Medical Oncology Hematology, Horsham, Pennsylvania
  - SCRI - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology Medical City Dallas, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - UT Health Science Center, Houston, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - VA Puget Sound, Seattle, Washington
- Australia (9):
  - Northern Cancer Insitute, St. Leonards, Saint Leonards, New South Wales
  - Royal Hobart Hospital, Hobart, Tasmania
  - Peninsula & Southeast Oncology, Frankston, Victoria
  - Barwon Health, University Hospital Geelong, Geelong, Victoria
  - Cabrini Hospital, Malvern, Victoria
  - Southside Cancer Care Centre, Miranda
  - Orange Health Services, Orange
  - St John of God Hospital, Subiaco, Subiaco
  - Riverina Cancer Care Centre, Wagga Wagga
- Belgium (6):
  - ZNA Middelheim, Antwerp
  - Universitair Ziekenhuis Gent, Ghent
  - AZ Groeninge, Kortrijk
  - CHU Sart-Tilman, Liège
  - Equipe de Recherche Clinique, Département d'Oncologie/Hématologie, Liège
  - AZ DELTA, Roeselare
- Canada (4):
  - Juravinski Cancer Centre Hamilton Health Services, Hamilton, Ontario
  - London Health Science Center - Victoria Hospital, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto
- Denmark (3):
  - Copenhagen University Hospital, Copenhagen
  - Herlev Hospital, Herlev
  - Vejle Sygehus, Vejle
- France (8):
  - Centre François Baclesse, Caen
  - Centre Georges François Leclerc, Dijon
  - Clinique Victor Hugo Centre Jean Bernard, Le Mans
  - Hôpital Privé La Louvière, Lille
  - Polyclinique de Gentilly (Centre D'Oncologie De Gentilly), Nancy
  - Institut Curie, Paris
  - Hôpital Privé des Côtes d'Armor, Plérin
  - CRLCC Eugene Marquis, Rennes
- Germany (14):
  - Gemeinschaftspraxis fur Hamatologie & Onkologie, Augsburg
  - Charite Universitatsmedizin Berlin, Berlin
  - Universitätsklinik Köln, Cologne
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - Universitatsklinikum Dusseldorf, Düsseldorf
  - Urologische Gemeinschaftspraxis, Emmendingen
  - Universitaetsklinikum Hamburg-Eppendorf (UKE), Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitatsklinikum Jena, Jena
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Medizinischen Fakultät Mannheim der Universität Heidelberg, Mannheim
  - Studienpraxis Urologie, Nürtingen
  - University of Tuebingen, Tübingen
  - Die Gesundhehitsunion DGU, Wuppertal
- Ireland (5):
  - Cork University Hospital, Cork
  - St. Vincent's University Hospital, Dublin
  - St James's Hospital, Dublin
  - Adelaide & Meath Hospital, Incorporating the National Children's Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
- Israel (6):
  - Rambam Health Care Campus (RHCC), Rambam Medical Center, Haifa
  - Hadassah University Hospital, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - The Tel Aviv Sourasky Medical Center (Ichilov Hospital), Tel Aviv
- Italy (8):
  - Ospedale San Donato, Azienda USLSUDEST, Arezzo
  - Ospedale Santa Maria delle Croci, Faenza
  - IRCCS Istituto Nazionale dei Tumori (INT), Milan
  - IEO Instituto Europeo di Oncologia, Milan
  - University of Modena and Reggio Emilia Medical Oncology, Modena
  - Azienda Ospedaliera San Camillo-Forlanini, Rome
  - Azienda Opsedaliera S. Maria di Terni, Terni
  - Santa Chiara Hospital, Dept Medical Oncology, Trento
- Spain (17):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital del Mar, Servicio de Oncología, Barcelona
  - Hospital Clínic i Provincial de Barcelona-Oncology, Barcelona
  - Instituto Catalan de Oncologia, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital General Universitario de Guadalajara, Guadalajara
  - Hospital Universitario Lucus Augusti., Lugo
  - MD Anderson Cancer Center - Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Puerta de Hierro-Majadahonda, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Corporacio Sanitaria Parc Tauli, Sabadell
  - Marques de Valdecilla University Hospital (HUMV), Santander
  - Hospital Universitario Virgen del Rocío, Seville
  - Instituto Valenciano de Oncologia IVO, Valencia
- United Kingdom (11):
  - Wexham Park Hospital, Slough, Berkshire
  - Mount Vernon Cancer Centre, Northwood, England
  - Royal Marsden Hospital, Sutton, Surrey
  - Oxford University Hospitals, Headington
  - Royal Liverpool Hospital, Liverpool
  - London Health Science Center - Victoria Hospital, London
  - Guy's Hospital, London
  - Sarah Cannon Research Institutute - UK, London
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral
  - Southampton General Hospital, Southampton
  - Musgrove Park Hospital, Taunton

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets for study results will be made available to qualified researchers in compliance with applicable privacy laws and data protection regulations.
  Data will be provided by Clovis Oncology.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available to qualified researchers after the primary, secondary, and/or exploratory outcomes of the study are reported or published and for 1 year thereafter.
Access Criteria: Requests for de-identified datasets will be made available to qualified researchers following submission of a methodologically sound proposal to medinfo@clovisoncology.com.

REFERENCES:
- [Derived] Abida W, Campbell D, Patnaik A, Bryce AH, Shapiro J, Bambury RM, Zhang J, Burke JM, Castellano D, Font A, Ganju V, Hardy-Bessard AC, McDermott R, Sautois B, Spaeth D, Voog E, Piulats JM, Pintus E, Ryan CJ, Merseburger AS, Daugaard G, Heidenreich A, Fizazi K, Loehr A, Despain D, Simmons AD, Dowson M, Go J, Watkins SP, Chowdhury S. Rucaparib for the Treatment of Metastatic Castration-resistant Prostate Cancer Associated with a DNA Damage Repair Gene Alteration: Final Results from the Phase 2 TRITON2 Study. Eur Urol. 2023 Sep;84(3):321-330. doi: 10.1016/j.eururo.2023.05.021. Epub 2023 Jun 3. PMID 37277275
- [Derived] Collins K, Cheng L. Reprint of: morphologic spectrum of treatment-related changes in prostate tissue and prostate cancer: an updated review. Hum Pathol. 2023 Mar;133:92-101. doi: 10.1016/j.humpath.2023.02.007. Epub 2023 Mar 8. PMID 36898948
- [Derived] Green ML, Ma SC, Goble S, Giordano H, Maloney L, Simmons AD, Beltman J, Harding TC, Xiao JJ. Population pharmacokinetics of rucaparib in patients with advanced ovarian cancer or other solid tumors. Cancer Chemother Pharmacol. 2022 May;89(5):671-682. doi: 10.1007/s00280-022-04413-7. Epub 2022 Apr 10. PMID 35397664
- [Derived] Maia MC, Salgia M, Pal SK. Harnessing cell-free DNA: plasma circulating tumour DNA for liquid biopsy in genitourinary cancers. Nat Rev Urol. 2020 May;17(5):271-291. doi: 10.1038/s41585-020-0297-9. Epub 2020 Mar 17. PMID 32203306

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 277 patients were recruited from 102 sites across 12 countries.
Groups:
- BRCA Mutation: Patients with a deleterious BRCA (breast cancer susceptibility gene) mutation detected in their tumor.
- ATM Mutation: Patients with a deleterious ATM (ataxia telangiectasia mutated serine/threonine kinase) mutation detected in their tumor.
- CDK12 Mutation: Patients with a deleterious CDK12 (Cyclin-dependent kinase 12) mutation detected in their tumor.
- CHEK2 Mutation: Patients with a deleterious CHEK2 (Checkpoint Kinase 2) mutation detected in their tumor.
- Other Gene Mutation: Patients with other deleterious HRR (homologous recombination repair) gene mutation detected in their tumor.
Period: Overall Study
Arm/Group | BRCA Mutation | ATM Mutation | CDK12 Mutation | CHEK2 Mutation | Other Gene Mutation
Started | 172 | 59 | 14 | 7 | 25
Completed | 172 | 59 | 14 | 7 | 25
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BRCA Mutation | ATM Mutation | CDK12 Mutation | CHEK2 Mutation | Other Gene Mutation | Total
Number analyzed (Participants) | 172 | 59 | 14 | 7 | 25 | 277
Age, Continuous [Median (Full Range); unit: years] | 72 [49 to 88] | 73 [51 to 84] | 64 [49 to 79] | 65 [60 to 86] | 70 [57 to 83] | 71 [49 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 172 | 59 | 14 | 7 | 25 | 277
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 0 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 8 | 3 | 1 | 0 | 4 | 16
  White | 127 | 43 | 6 | 5 | 17 | 198
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 33 | 13 | 7 | 1 | 3 | 57

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Response Rate (ORR) by Gene in Patients With Measurable Disease at Baseline Per Central Independent Radiology Review (IRR)
Description: The primary efficacy endpoint is confirmed radiographic ORR by central IRR. ORR is defined as the percentage of patients with a confirmed CR (complete response) or PR (partial response) by mRECIST (modified Response Evaluation Criteria in Solid Tumors) v1.1/PCWG3 (Prostate Cancer Working Group 3) criteria. The confirmed response is defined as a CR or PR on subsequent tumor assessment at least 28 days after first response documentation in the absence of confirmed progression in bone. CR is disappearance of all target and non-target lesions; any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Assessments every 8 weeks from study day 1 for the first 24 weeks, and then every 12 weeks until disease progression, death, or initiation of subsequent treatment. Total follow-up was up to approximately 3 years.
Population: IRR Efficacy Population - The IRR efficacy population is defined by measurable disease status at baseline using modified RECIST Version 1.1 criteria per independent radiology review.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BRCA Mutation | ATM Mutation | CDK12 Mutation | CHEK2 Mutation | Other Gene Mutation
Number analyzed (Participants) | 81 | 23 | 8 | 4 | 17
percentage of participants | 45.7 [34.6 to 57.1] | 0.0 [0.0 to 14.8] | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 60.2] | 41.2 [18.4 to 67.1]

2. Secondary Outcome: Confirmed Objective Response Rate (ORR) by Gene in Patients With Measurable Disease at Baseline Per Investigator (INV)
Description: A supportive efficacy endpoint is confirmed radiographic ORR by INV. ORR is defined as the percentage of patients with a confirmed CR (complete response) or PR (partial response) by mRECIST (modified Response Evaluation Criteria in Solid Tumors) v1.1/PCWG3 (Prostate Cancer Working Group 3) criteria. The confirmed response is defined as a CR or PR on subsequent tumor assessment at least 28 days after first response documentation in the absence of confirmed progression in bone. CR is disappearance of all target and non-target lesions; any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: as for outcome 1
Population: Investigator Efficacy Population - The Investigator efficacy population is defined by measurable disease status at baseline using modified RECIST Version 1.1 criteria per the investigator (INV).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BRCA Mutation | ATM Mutation | CDK12 Mutation | CHEK2 Mutation | Other Gene Mutation
Number analyzed (Participants) | 87 | 21 | 9 | 4 | 17
percentage of participants | 48.3 [37.4 to 59.2] | 9.5 [1.2 to 30.4] | 0.0 [0.0 to 33.6] | 25.0 [0.6 to 80.6] | 41.2 [18.4 to 67.1]

3. Secondary Outcome: Duration of Response (DOR) by Gene in Patients With Confirmed Response Per Central Independent Radiology Review (IRR)
Description: A secondary efficacy endpoint is DOR by central IRR. The DOR is defined as the time from the date that a confirmed response per modified RECIST Version 1.1/PCWG3 is first reported to the time that progressive disease (PD) is first documented. Progressive disease is defined using RECIST v1.1, as at least a 20% increase in the sum of the diameters of target lesions, or an unequivocal increase in non-target lesions, or the appearance of new lesions. PCWG3 criteria is used to document evidence of disease progression in bone lesions.
Time Frame: as for outcome 1
Population: Patients with a confirmed response in the IRR Efficacy Population. The IRR efficacy population is defined by measurable disease status at baseline using modified RECIST Version 1.1 criteria per independent radiology review. Note, there were no patients with confirmed response by IRR in the ATM, CDK12 and CHEK2 arms.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BRCA Mutation | Other Gene Mutation
Number analyzed (Participants) | 37 | 7
months | 15.5 [6.4 to NA] — The upper confidence interval was not assessable due to insufficient number of participants with events. | 22.1 [10.1 to NA] — The upper confidence interval was not assessable due to insufficient number of participants with events.

4. Secondary Outcome: Duration of Response (DOR) by Gene in Patients With Confirmed Response Per Investigator
Description: A secondary efficacy endpoint is DOR as assessed by the investigator. The DOR is defined as the time from the date that a confirmed response per modified RECIST Version 1.1/PCWG3 is first reported to the time that progressive disease (PD) is first documented. Progressive disease is defined using RECIST v1.1, as at least a 20% increase in the sum of the diameters of target lesions, or an unequivocal increase in non-target lesions, or the appearance of new lesions. PCWG3 criteria is used to document evidence of disease progression in bone lesions.
Time Frame: as for outcome 1
Population: Patients with a confirmed response in the Investigator Efficacy Population. The Investigator efficacy population is defined by measurable disease status at baseline using modified RECIST Version 1.1 criteria per the investigator. Note, there were no patients with confirmed response by investigator in the CDK12 arm.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BRCA Mutation | ATM Mutation | CHEK2 Mutation | Other Gene Mutation
Number analyzed (Participants) | 42 | 2 | 1 | 7
months | 6.6 [5.6 to 11.6] | 7.5 [4.6 to 10.4] | 16.6 [NA to NA] — The median is the actual observed value for this participant. The confidence interval was not assessable due to insufficient number of participants with events. | 18.4 [10.1 to NA] — The upper confidence interval was not assessable due to insufficient number of participants with events.

5. Secondary Outcome: Confirmed PSA Response (≥ 50% Decrease) by Gene as Assessed by Local Laboratory
Description: A secondary endpoint is confirmed PSA (prostate-specific antigen) response (≥ 50% reduction) as assessed by local laboratory. Confirmed PSA response is analyzed for all patients who had PSA value at baseline and is defined as the percentage of patients having 2 consecutive PSA values (at least 3 weeks apart) that are at least 50% lower than baseline and that occur prior to PSA progression. PSA progression is defined as a ≥ 25% increase and absolute increase of ≥ 2 ng/mL above the nadir in PSA.
Time Frame: PSA assessments were done at baseline, Week 5, Week 9, every 4 weeks thereafter, and at Treatment Discontinuation. Total follow-up was up to approximately 39 months.
Population: All patients who had a PSA value at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BRCA Mutation | ATM Mutation | CDK12 Mutation | CHEK2 Mutation | Other Gene Mutation
Number analyzed (Participants) | 172 | 59 | 14 | 7 | 25
percentage of participants | 53.5 [45.7 to 61.1] | 3.4 [0.4 to 11.7] | 7.1 [0.2 to 33.9] | 14.3 [0.4 to 57.9] | 36.0 [18.0 to 57.5]

6. Secondary Outcome: Confirmed PSA Response (≥ 90% Decrease) by Gene as Assessed by Local Laboratory
Description: A secondary endpoint is confirmed PSA (prostate-specific antigen) response (≥ 90% reduction) as assessed by local laboratory. Confirmed PSA response is analyzed for all patients who had PSA value at baseline and is defined as the percentage of patients having 2 consecutive PSA values (at least 3 weeks apart) that are at least 90% lower than baseline and that occur prior to PSA progression. PSA progression is defined as a ≥ 25% increase and absolute increase of ≥ 2 ng/mL above the nadir in PSA.
Time Frame: as for outcome 5
Population: All patients who had a PSA value at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BRCA Mutation | ATM Mutation | CDK12 Mutation | CHEK2 Mutation | Other Gene Mutation
Number analyzed (Participants) | 172 | 59 | 14 | 7 | 25
percentage of participants | 19.8 [14.1 to 26.5] | 0 [0 to 0] | 0 [0 to 0] | 14.3 [0.4 to 57.9] | 16.0 [4.5 to 36.1]

7. Secondary Outcome: Radiologic Progression-free Survival (rPFS) by Gene in All Patients Per Central Independent Radiology Review (IRR)
Description: A secondary efficacy endpoint is Radiologic Progression-free Survival (rPFS) assessed by IRR. rPFS is defined as the time from first dose of rucaparib to the date of first objective evidence of radiographic progression (soft tissue or bone lesion) or death due to any cause, whichever occurs first, plus 1 day. Radiographic disease progression includes confirmed bone disease progression and soft tissue disease progression adjudicated by IRR using the PCWG3 guidelines for bone disease and modified RECIST Version 1.1 for soft tissue disease.
Time Frame: as for outcome 1
Population: All patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BRCA Mutation | ATM Mutation | CDK12 Mutation | CHEK2 Mutation | Other Gene Mutation
Number analyzed (Participants) | 172 | 59 | 14 | 7 | 25
months | 10.7 [8.7 to 13.2] | 5.3 [3.7 to 8.9] | 3.7 [1.9 to 8.3] | 9.4 [2.1 to NA] — The upper confidence interval was not assessable due to insufficient number of participants with events. | 11.6 [5.1 to 25.3]

8. Secondary Outcome: Radiologic Progression-free Survival (rPFS) by Gene in All Patients Per Investigator
Description: A secondary efficacy endpoint is Radiologic Progression-free Survival (rPFS) assessed by Investigator. rPFS is defined as the time from first dose of rucaparib to the date of first objective evidence of radiographic progression (soft tissue or bone lesion) or death due to any cause, whichever occurs first, plus 1 day. Radiographic disease progression includes confirmed bone disease progression and soft tissue disease progression using the PCWG3 guidelines for bone disease and modified RECIST Version 1.1 for soft tissue disease.
Time Frame: as for outcome 1
Population: All patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BRCA Mutation | ATM Mutation | CDK12 Mutation | CHEK2 Mutation | Other Gene Mutation
Number analyzed (Participants) | 172 | 59 | 14 | 7 | 25
months | 9.6 [8.2 to 11.2] | 7.8 [4.2 to 10.6] | 3.7 [1.9 to 8.1] | 3.5 [2.1 to 11.2] | 11.6 [5.8 to 22.3]

9. Secondary Outcome: Overall Survival (OS) by Gene
Description: A secondary efficacy endpoint is Overall Survival (OS). OS is defined as the date from first dose of rucaparib to the date of death due to any cause, +1 day.
Time Frame: From date of first dose until event, loss to follow-up, withdrawal of consent, or study closure: an overall median of approximately 33.1 months
Population: Safety Population - The safety population consists of all patients who received at least 1 dose of protocol-specified treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BRCA Mutation | ATM Mutation | CDK12 Mutation | CHEK2 Mutation | Other Gene Mutation
Number analyzed (Participants) | 172 | 59 | 14 | 7 | 25
months | 17.2 [14.8 to 20.0] | 14.6 [12.0 to 19.0] | 13.9 [6.8 to 18.6] | 11.1 [3.5 to 26.7] | 11.6 [8.9 to NA] — The upper confidence interval was not assessable due to insufficient number of participants with events.

10. Secondary Outcome: Clinical Benefit Rate (CBR) by Gene Per Central Independent Radiology Review (IRR)
Description: A secondary efficacy endpoint is Clinical Benefit Rate (CBR) assessed by IRR. CBR is defined as the number of patients without radiographic progression (defined by modified RECIST Version 1.1/ PCWG3 criteria) who were continuing with study drug treatment through the given time interval divided by the number of patients who had the given amount of follow-up. Clinical benefit rates are summarized at 6 and 12 months.
Time Frame: as for outcome 1
Population: All patients
Measure: Count of Participants; unit: Participants
Arm/Group | BRCA Mutation | ATM Mutation | CDK12 Mutation | CHEK2 Mutation | Other Gene Mutation
Number analyzed (Participants) | 172 | 59 | 14 | 7 | 25
Participants
  6 months | 100 | 10 | 2 | 2 | 13
  12 months | 36 | 3 | 0 | 1 | 6

11. Secondary Outcome: Clinical Benefit Rate (CBR) by Gene Per Investigator
Description: A secondary efficacy endpoint is Clinical Benefit Rate (CBR) assessed by Investigator. CBR is defined as the number of patients without radiographic progression (defined by modified RECIST Version 1.1/ PCWG3 criteria) who were continuing with study drug treatment through the given time interval divided by the number of patients who had the given amount of follow-up. Clinical benefit rates are summarized at 6 and 12 months.
Time Frame: as for outcome 1
Population: All patients
Measure: Count of Participants; unit: Participants
Arm/Group | BRCA Mutation | ATM Mutation | CDK12 Mutation | CHEK2 Mutation | Other Gene Mutation
Number analyzed (Participants) | 172 | 59 | 14 | 7 | 25
Participants
  6 months | 103 | 17 | 3 | 2 | 14
  12 months | 39 | 6 | 1 | 1 | 6

12. Secondary Outcome: Time to PSA Progression by Gene
Description: A secondary efficacy endpoint is time to PSA progession. Time to PSA progression is defined as the time from first dose of rucaparib to the date that a ≥ 25% increase and absolute increase of ≥ 2 ng/mL above the nadir (or baseline if there was no PSA decline after baseline) in PSA was measured, plus 1 day. The increase must be confirmed by a second consecutive assessment conducted at least 3 weeks later (unless the PSA progression occurred at the last recorded PSA assessment). If confirmed, the date used for time of PSA progression is the earlier of the 2 PSA dates.
Time Frame: as for outcome 5
Population: All patients who had a PSA value at baseline.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BRCA Mutation | ATM Mutation | CDK12 Mutation | CHEK2 Mutation | Other Gene Mutation
Number analyzed (Participants) | 172 | 59 | 14 | 7 | 25
months | 6.5 [5.7 to 7.5] | 3.1 [2.8 to 3.7] | 3.5 [2.8 to 4.6] | 5.6 [2.8 to NA] — The upper confidence interval was not assessable due to insufficient number of participants with events. | 5.3 [3.0 to 9.1]

13. Secondary Outcome: Steady State Trough (Cmin) Level Rucaparib Concentrations
Description: Trough (Cmin) concentrations of rucaparib are summarized for all patients with at least one PK sample collected. The absolute values of rucaparib plasma concentration at each time point are presented by gene.
Time Frame: Participants were assessed at Study Day 29, Day 57, Day 85 and Day 113
Population: Safety population with at least one PK sample collected. The safety population consists of all patients who received at least 1 dose of protocol-specified treatment.
Measure: Median (Standard Deviation); unit: ng/mL
Arm/Group | BRCA Mutation | ATM Mutation | CDK12 Mutation | CHEK2 Mutation | Other Gene Mutation
Number analyzed (Participants) | 101 | 51 | 14 | 5 | 13
ng/mL
  Day 29: number analyzed (Participants) | 101 | 48 | 14 | 5 | 13
  Day 29 | 1539.565 (966.2604) | 1605.002 (856.2478) | 1639.357 (1428.5691) | 1286.998 (1138.2119) | 1189.845 (748.3045)
  Day 57: number analyzed (Participants) | 85 | 38 | 12 | 3 | 11
  Day 57 | 1578.353 (1057.8049) | 1600.380 (1198.3899) | 1405.167 (806.4642) | 1841.667 (2106.3362) | 1792.499 (1672.7732)
  Day 85: number analyzed (Participants) | 71 | 30 | 10 | 2 | 9
  Day 85 | 1308.704 (693.6717) | 1505.400 (802.0812) | 1699.700 (991.9922) | 815.500 (557.9073) | 2255.889 (1831.9626)
  Day 113: number analyzed (Participants) | 60 | 22 | 10 | 2 | 8
  Day 113 | 1533.690 (889.6130) | 1515.300 (1291.8497) | 1520.700 (884.1374) | 728.000 (469.5189) | 1433.875 (637.4535)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from date of first dose of study drug until 28 days after last dose of study drug, approximately 4.5 years.
Groups:
- All Patients: All patients received open-label oral rucaparib 600 mg BID (twice a day) in continuous 28-day cycles.
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 8/277
Serious Adverse Events (participants affected / at risk) | 96/277
Other Adverse Events (participants affected / at risk) | 274/277
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=277)
Anaemia (Blood and lymphatic system disorders) | 14
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1
Aplastic anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 2
Acute coronary syndrome (Cardiac disorders) | 3
Acute myocardial infarction (Cardiac disorders) | 3
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Coronary artery occlusion (Cardiac disorders) | 1
Torsade de pointes (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1
Mechanical ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Oesophagitis (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 2
Fatigue (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 2
Pyrexia (General disorders) | 1
Abscess oral (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 2
Fournier's gangrene (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Haemophilus infection (Infections and infestations) | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2
Legionella infection (Infections and infestations) | 1
Paraspinal abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 6
Pneumonia legionella (Infections and infestations) | 1
Pneumonia staphylococcal (Infections and infestations) | 1
Pulmonary sepsis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 4
Urosepsis (Infections and infestations) | 4
Wound infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 2
Foot fracture (Injury, poisoning and procedural complications) | 1
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 5
Spinal pain (Musculoskeletal and connective tissue disorders) | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebellar infarction (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Sacral radiculopathy (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 2
Spinal cord compression (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Confusional state (Psychiatric disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 7
Haematuria (Renal and urinary disorders) | 6
Hydronephrosis (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Embolism (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=277)
Anaemia (Blood and lymphatic system disorders) | 129
Neutropenia (Blood and lymphatic system disorders) | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 33
Abdominal pain (Gastrointestinal disorders) | 16
Constipation (Gastrointestinal disorders) | 76
Diarrhoea (Gastrointestinal disorders) | 65
Dyspepsia (Gastrointestinal disorders) | 18
Nausea (Gastrointestinal disorders) | 139
Vomiting (Gastrointestinal disorders) | 67
Asthenia (General disorders) | 50
Fatigue (General disorders) | 131
Oedema peripheral (General disorders) | 50
Pyrexia (General disorders) | 15
Upper respiratory tract infection (Infections and infestations) | 19
Urinary tract infection (Infections and infestations) | 37
Fall (Injury, poisoning and procedural complications) | 18
Alanine aminotransferase increased (Investigations) | 72
Aspartate aminotransferase increased (Investigations) | 71
Blood alkaline phosphatase increased (Investigations) | 18
Blood creatinine increased (Investigations) | 50
Platelet count decreased (Investigations) | 32
Weight decreased (Investigations) | 45
Decreased appetite (Metabolism and nutrition disorders) | 96
Dehydration (Metabolism and nutrition disorders) | 14
Hypocalcaemia (Metabolism and nutrition disorders) | 21
Hypophosphataemia (Metabolism and nutrition disorders) | 27
Althralgia (Musculoskeletal and connective tissue disorders) | 44
Back pain (Musculoskeletal and connective tissue disorders) | 50
Bone pain (Musculoskeletal and connective tissue disorders) | 18
Muscular weakness (Musculoskeletal and connective tissue disorders) | 17
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 14
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 33
Myalgia (Musculoskeletal and connective tissue disorders) | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 32
Dizziness (Nervous system disorders) | 53
Dysgeusia (Nervous system disorders) | 32
Headache (Nervous system disorders) | 28
Neuropathy peripheral (Nervous system disorders) | 14
Insomnia (Psychiatric disorders) | 18
Haematuria (Renal and urinary disorders) | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 40
Dry skin (Skin and subcutaneous tissue disorders) | 18
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 19
Rash (Skin and subcutaneous tissue disorders) | 22
Hypertension (Vascular disorders) | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor's agreements with investigators require proposed public disclosures of trial results to be submitted to Sponsor for review prior to publication. Sponsor may request deletion of confidential information or a delay in publication to address intellectual property concerns, but Sponsor may not suppress publication of the trial results indefinitely. Sponsor may request delay of a single-center publication until after the release of a multi-site publication or an agreed upon period of time.

DOCUMENTS (2):
  • Study Protocol (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/34/NCT02952534/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT02952534/SAP_001.pdf